CLINICAL TRIAL: NCT04717154
Title: Phase 2 INSPIRE Trial: Ipilimumab With Nivolumab for Molecular- Selected Patients With Castration-resistant Prostate Cancer
Brief Title: Ipilimumab With Nivolumab for Molecular-selected Patients With Castration-resistant Prostate Cancer
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOURO048 - INSPIRE; 2020-001240-25 (EudraCT Number); CA184-585 (Other: Bristol Meyers Squibb)
Record Dates: First submitted 2021-01-06; First posted 2021-01-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-04

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: mCRPC; Immune checkpoint inhibitors; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Intervention Model Description: Open label, single treatment, phase II study:
  * Cohort A1 will assess the efficacy of ipilimumab+nivolumab in mCRPC patients with RECIST1.1 measurable disease that are naïve for immune checkpoint inhibition
  * Cohort A2 will assess the efficacy of ipilimumab+nivolumab in patients without RECIST1.1 measurable disease that are naïve for immune checkpoint inhibition
  * Cohort B will assess the efficacy of ipilimumab+nivolumab in patients with RECIST1.1 measurable disease and prior progression to immune checkpoint inhibitor monotherapy (CTLA-4 or anti-PD1/PDL1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Combinatory regimen of nivolumab 3mg/kg and ipilimumab 1mg/kg, followed by nivolumab 480mg flat dose (Q4w) to up to one year.
  This regimen will be given to participants in both cohort 1 and 2.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — 4 courses of 1mg/kg q3w
  Other Names: Yervoy, BMS-734016, MDXOIO, MDX-CTLA4
Biological: Nivolumab — 4 courses of 3mg/kg q3w, followed by maintenance flat dose (480mg, q4w, for 10 doses)
  Other Names: Opdivo, BMS-936558, MDX1106, ONO-4538

SUMMARY:
The purpose of this study is to evaluate the effects of 4 cycles of combinatory immunotherapy (ipilimumab and nivolumab), followed by monotherapy nivolumab in participants with immunogenic metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Following molecular characterization (next-generation sequencing) a total of 75 mCRPC patients with a putative immunogenic subtype will be included within the phase 2 INSPIRE trial. As treatment we will be utilizing a combinatory regimen of nivolumab 3mg/kg and ipilimumab 1mg/kg for 4 doses, followed by nivolumab 480mg flat dose for up to one year. All participants will additionally undergo an on-trial metastatic tissue biopsy. Translational research will study immunological correlates and in-depth genomic/transcriptomic and multispectral immunohistochemical analyses of immune infiltrate.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Written informed consent.
2. Histological diagnosis of adenocarcinoma of the prostate. Patients who have no histological diagnosis must be willing to undergo a biopsy to prove prostate adenocarcinoma.
3. Metastatic Castration-Resistant Prostate Cancer (mCRPC), metastatic disease defined either as measurable disease by RECIST1.1 criteria or presence of bone-metastatic disease evaluable per PCWG3 criteria. For cohort 1, measurable disease is compulsory.
4. An immunogenic phenotype, consisting of one of the next criteria: 1, mismatch repair deficiency and/or a high mutational burden of >7 mutations per Mb (cluster A); 2, BRCA2 inactivation or BRCAness signature (cluster B); 3, a tandem duplication signature and/or CDK12 biallelic inactivation (cluster C)
5. Age ≥18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
7. PSA ≥ 2 ng/ml.
8. Documented willingness to use an effective means of contraception while participating in the study and for 7 months post last dose of treatment
9. Documented ongoing castrate serum testosterone <50 ng/dL (<2.0 nM).
10. Received prior castration by orchiectomy and/or ongoing Luteinizing Hormone-Releasing Hormone (LH-RH) agonist treatment.
11. Progression of disease by:

    1. PSA utilizing PCWG3 criteria
    2. Bone scan: disease progression as defined by at least 2 new lesions on bone scan.
    3. Soft tissue disease progression defined by modified RECIST 1.1.
    4. Clinical progression with worsening pain and the need for palliative radiotherapy for bone metastases.
12. Having a biopsiable metastatic lesion and willingness to undergo a baseline* and on treatment tumour biopsy for next-generation sequencing and biomarker analyses.

    * When sufficient FFPE material is available from a biopsy in castrate-state, one may apply for a waiver for a new baseline biopsy.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Prior treatment with checkpoint immunotherapy (CTLA-4, or PD-1 and PD-L1 antagonists) for cohort 1. For cohort 2, patients may have prior treatment with monotherapy CTLA-4 or PD-1 or PD-L1.
2. Surgery or chemotherapy within 4 weeks prior to trial entry / randomisation into the study. Any other therapies for prostate cancer, other than GnRH analogue therapy and osteoporosis preventing agents, are not allowed.
3. Radiotherapy within 2 weeks prior to trial entry. Radiation-related side effects higher than grade 1, or above baseline.
4. Participation in another interventional clinical trial and any concurrent treatment with any investigational drug within 4 weeks prior to trial entry/randomisation.
5. History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumours, brain metastases, or alcoholism.
6. Untreated or symptomatic brain or leptomeningeal involvement.
7. Inadequate organ and bone marrow function as evidenced by:

   1. hemoglobin <6.2 mmol/L
   2. Absolute neutrophil count <1.0 x 109/L
   3. Platelet count < 75 x 109/L
   4. Albumin <30 g/dL.
   5. AST / SGOT and/or ALT / SGPT ≥ 2.5 x ULN (≥ 5 x ULN if liver metastases present)
   6. Total bilirubin ≥ 1.5 x ULN (except for patient with documented Gilbert's disease)
   7. Serum Creatinine > 1.5 x ULN
8. Any of the following cardiac criteria; a. Any clinically significant abnormalities in rhythm conduction, or morphology of a resting ECG (e.g., complete left bundle branch block, third degree heart block) c. Experience of any of the following procedures or conditions in the preceding six months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, congestive heart failure NYHA ≥ Grade2 d. Uncontrolled hypotension defined as systolic blood pressure (BP) <90mmHg and/or diastolic BP <50mmHg
9. Clinically significant history of liver disease consistent with Child-Pugh Class B or C, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
10. History of clinically relevant auto-immune disease (including Crohn's disease or ulcerative colitis). Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of nivolumab or ipilimumab or that may affect the interpretation of the results or renders the patients at high risk from treatment complications.
11. Need for chronic corticosteroid therapy of >10 mg of prednisolone or >0.5mg of dexamethasone per day or an equivalent dose of other anti-inflammatory corticosteroid. Patients in which corticosteroids cannot be stopped prior to entering the trial are allowed a maximum of 10mg of prednisolone per day or equivalent. In the case of corticosteroid discontinuation, a 2-week (14 days) washout is required with a mandatory PSA check prior to starting the trial. If the PSA has declined compared to the value obtained prior to stopping corticosteroids, patients will not be eligible for study. Patients can only enter the study with a confirmed PSA increase.
12. Malignancies other than prostate cancer within 3 years prior to trial entry / randomization, except for adequately treated basal or squamous cell skin cancer and non-muscle invasive bladder cancer.
13. Active second malignancy, except basal or squamous cell skin cancer and non-muscle invasive bladder cancer. Other treated malignancies with curative intent, including colorectal cancer, may be included following PI consent.
14. Unresolved clinically significant toxicity from prior therapy except for alopecia and Grade 1 peripheral neuropathy.
15. Inability to comply with study and follow-up procedures.
16. Patients with predominant small cell or neuroendocrine prostate cancer are not eligible.
17. Patients without measurable lesion per RECIST1.1, and with a superscan on bone scintigraphy not evaluable per PCWG3 criteria, are not eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint: DCR | At inclusion, Weeks 7, 17, 29, and 41, and 30 days after last dose given at week 49
  For patients with RECIST1.1 evaluable disease this includes a change from baseline in tumour volume as measured by PR or CR by best ORR, or an SD, all lasting longer than 6mo, and the absence of clinical disease progression.
  In patients without RECIST1.1 evaluable disease, disease control is defined by the absence of new measurable lesions and unequivocal PD of non-target lesions on CT scan, the absence of bone progression as defined by the PCWG3 criteria, and the absence of clinical disease progression

SECONDARY OUTCOMES:
Safety endpoint: adverse effects | At inclusion, Weeks 1, 4, 7, 10, 13, 17, 21, 25, 29, 33, 37, 41, 45, and 49, and at end of treatment (typically at one year, or earlier when treatment is stopped prematurely)
  Percentage of Grade 3/4 and 5 treatment-related adverse effects
Efficacy endpoint: ORR | At inclusion, Weeks 7, 17, 29, and 41, and 30 days after last dose given at week 49
  Best objective response rate (ORR) per RECIST1.1 criteria (cohort A1 only)
Efficacy endpoint: BRR | BRR at Week 13, PSA at inclusion, Weeks 1, 4, 7, 10, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49 and at end of treatment (typically one year, or earlier when treatment is stopped prematurely)
  Biochemical response rate (BRR) at week 13 and maximal PSA decline according to PCWG3 criteria
Efficacy endpoint: rPFS | At inclusion, Weeks 7, 17, 29, and 41, and 30 days after last dose given at week 49
  Radiographic progression free survival per irRECIST1.1 immune-related response criteria
Efficacy endpoint: OS | Follow-up of 1 year following trial discontinuation (onwards from the 30-day safety follow-up visit).
  Overall survival
Efficacy in the BRCA, CDK12 and MSI/hTMB subgroups | At inclusion, Weeks 7, 17, 29, and 41, and 30 days after last dose given at week 49
  DCR, ORR, BRR, rPFS and OS per subgroup
Efficacy in the subgroup of patients with prior RT | At inclusion, Weeks 7, 17, 29, and 41, and 30 days after last dose given at week 49
  DCR, ORR, BRR, rPFS and OS in patients with and without prior radiotherapy

OTHER OUTCOMES:
Translational endpoint: biomarkers | Through study completion, an average of 2 years
  To further optimize and validate predictive and early response immunogenic signatures from biomarkers in tissue and blood, associating with an objective response and disease control (DCR) of at least 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Niven Mehra, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided